CLINICAL TRIAL: NCT02245334
Title: A Prospective Randomized Trial of Povidone-iodine Suppository Before Transrectal Ultrasound Guided Prostate Biopsy
Brief Title: A Prospective Trial of Povidone-iodine Suppository Before Transrectal Ultrasound Guided Prostate Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-1403/243-004
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Infection; Prostatic Diseases; Misadventure During Aspirating Needle Biopsy
MeSH Terms: conditions — Infections; Prostatic Diseases | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Povidone-iodine (Experimental): povidone iodine pill
  Interventions: Drug: Povidone-Iodine
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Drug: Povidone-Iodine — 1 pill per biopsy
  Other Names: Gynobetadine
  Arms: Povidone-iodine

SUMMARY:
To assess the effect of povidone-iodine on infectious complication rate caused by transrectal prostate biopsy

DETAILED DESCRIPTION:
the effect of povidone-iodine on infectious complication rate caused by transrectal prostate biopsy

ELIGIBILITY:
Inclusion Criteria:

* who undergo transrectal prostate biopsy

Exclusion Criteria:

* patients who refuse to be included, patients who have hypersensitivity to iodine, patients who have abnormal thyroid function, patients who do not visit follow-up, patients who have received prior radioactive-iodine therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1578 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with febrile infection | 1 week
  consider fever over 38 degree celsius or admission due to fever

SECONDARY OUTCOMES:
voiding questionnaire | 1-2 week
  check International Prostate Symptom Score (IPSS)
sexual function questionnaire | 1-2 week
  International Index of Erectile Function-5 (IIEF-5)
quality of life questionnaire | 1-2 week
  European Organization for Research and Treatment fo Cancer (EORTC) Quality of life Questionnaire (QLQ)-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sangchul Lee, MD.PhD., Principal Investigator — Prof
Locations (1):
- Department of Urology, Seoul National University Bundang Hospital, Seongnam, Gyunggi-do, South Korea